CLINICAL TRIAL: NCT02197286
Title: Vitamin-D Treatment Targeted to Hyperprolinemia-Associated Schizophrenia.
Brief Title: Targeted Vitamin D Treatment of Schizophrenia-Associated Hyperprolinemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Personnel changes at study site.
Sponsor: NYU Langone Health (Other)
Collaborators: Stanley Medical Research Institute (Other); Columbia University (Other)
Responsible Party: Principal Investigator, James D. Clelland, Research Assistant Professor, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S13-01127
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (cholecalciferol) (Experimental): Intervention: Capsules containing the active ingredient, cholecalciferol @ 4,000 international units (IU). One capsule daily, oral administration for 10 weeks.
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): Daily matching placebo gelatin capsule (also contains microcrystalline cellulose).
  Capsules are identical in size, color and taste to experimental drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — One capsule containing 4,000 IU of Cholecalciferol, per day
  Other Names: Other name: Vitamin D3; Trade name:Biotech Pharmacal, Inc: Vitamin D3-4,; 4,000 IU per day
  Arms: Vitamin D (cholecalciferol)
Drug: Placebo — Daily dose of a single gelatin placebo capsule.
  Arms: Placebo

SUMMARY:
A ten week, blinded trial of vitamin D vs. placebo in 80 patients with schizophrenia or schizoaffective disorder who have low blood levels of vitamin D and elevated blood levels of the amino acid proline. The aims of the study are to evaluate an anticipated clinical response to vitamin D supplementation including negative symptoms and cognitive deficits, evaluate safety of vitamin D supplementation for schizophrenia patients and evaluate the relationship of changes in plasma proline levels and efficacy outcomes.

DETAILED DESCRIPTION:
25-hydroxyvitamin D (vitD) insufficiency is associated with cognitive decline and has long-been considered important in schizophrenia susceptibility. VitD supplementation has been suggested for those at-risk, and recent studies have demonstrated that vitD insufficiency extends into both adolescent and adult schizophrenia.

The mechanism by which vitD deficits confers risk is unknown. However, vitD is a transcriptional regulator, and the investigators recently found that vitD significantly up-regulates PRODH gene expression. This is important because the highest known genetic risk of schizophrenia is conferred by hemizygous microdeletion of chromosome 22q11, to which PRODH maps. Furthermore, PRODH encodes proline oxidase, which catalyzes proline catabolism. Proline is a neuromodulator at glutamatergic synapses, and peripheral hyperprolinemia has been associated with learning and memory deficits and neurotransmitter dysregulation in animal models, and in humans, with decreased intelligence quotient (IQ), cognitive impairment, and schizoaffective disorder. The investigators recently found that >25% of schizophrenia patients were hyperprolinemic and hypothesized a causal relationship between vitD, proline elevation, and schizophrenia, such that vitD insufficiency causes decreased PRODH expression and hyperprolinemia. Measuring fasting plasma 25hydroxyvitD and proline in 64 patients and 90 controls, the investigators found that vitD insufficiency (<30ng/ml) was significantly associated with schizophrenia (OR:2.1, p=0.044), vitD levels were negatively correlated with proline (p=0.01), and vitD insufficient subjects had three times greater odds of hyperprolinemia (p=0.046). Moreover, they demonstrated that hyperprolinemia explains >37% of the association between vitD insufficiency and schizophrenia, signifying that vitD insufficiency increases schizophrenia risk, at least in part by elevating proline. These findings advocate that targeting schizophrenia-associated hyperprolinemia by alleviating vitD insufficiency, may improve symptoms including neurocognitive deficits.

The Specific Aims of this study are:

Aim 1) To Evaluate a clinical response to vitamin D3 (vitD3) treatment, targeting patients with both vitD insufficiency and hyperprolinemia.

Aim 2) To Evaluate the relationship between fasting plasma proline change, PRODH expression, and symptoms, for development of an efficacy biomarker.

The aims will be accomplished via a ten week, double-blind, placebo controlled trial, in which schizophrenia or schizoaffective disorder subjects who are both vitD insufficient and hyperprolinemic, will be randomized to vitD3 (4,000 international units (IU)/day n=40) or placebo (n=40) as an adjunct to their antipsychotics.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Recruitment

1. Male and Female, all racial/ethnic groups, aged 18-65 years.
2. Admission diagnosis of schizophrenia, schizophreniform disorder, or schizoaffective disorder.
3. Capability to give informed consent.

Inclusion Criteria for Randomization and Trial Entry

1. Fasting hyperprolinemia (defined as 2 standard deviations (SDs) above the gender-adjusted mean measured for historical controls: 203.3 micromolar (uM) for females and 327.6 uM for males).
2. 25(OH)D insufficiency (<30ng/ml).
3. Confirmed diagnosis of schizophreniform disorder, schizophrenia or schizoaffective disorder.

Exclusion Criteria:

Exclusion Criteria for Recruitment

1. Organic brain disorders.
2. Valproate treatment within 14 days, because of known proline up-regulatory effects.
3. Pregnant women or women of child-bearing potential, who are not surgically-sterile or who are not using appropriate methods of birth control.
4. Amino acid metabolism disorder diagnosis.
5. Hypercalcemia (>10.4mg/dL), hypercalciuria (>0.20mg/mg), hyperthyroidism (>65pg/ml) or history of renal stones, kidney disease, atherosclerosis, sarcoidosis, histoplasmosis and lymphoma.
6. Chart record of HIV positive status.
7. Treatment with clozapine, as this may reflect general treatment resistance.

Exclusion Criteria for Randomization and Trial Entry

1. Abnormal serum/ urine metabolic lab values suggesting hypercalcemia (serum Calcium >10.4mg/dL), hypercalciuria (urine calcium/urine creatinine >0.20 mg/mg), or hyperthyroidism (parathyroid hormone (PTH) > 65pg/ml).
2. Initiation of Valproate treatment.
3. Continued use of dietary supplementation, such as fish oil supplementation or vitamin D supplements (>400 IU/day).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Clinical response to supplementation with vitamin D. | Baseline (start of vitamin D supplementation) through ten weeks of treatment.
  To evaluate an anticipated clinical response to supplementation with vitamin D including negative symptoms and cognitive deficits by the change in the Positive and Negative Symptom Scale (PANSS) total score and the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) consensus cognitive scale. Secondary outcomes will also involve investigation of individual domains of the PANSS and MATRICS.

SECONDARY OUTCOMES:
Biological response to supplementation with vitamin D. | Lead-in phase visit, baseline visit and then at biweekly visits through ten weeks of treatment.
  Measure plasma proline levels and peripheral PRODH gene expression levels, and examine the relationship with clinical symptoms and cognitive deficits for efficacy biomarker development.

OTHER OUTCOMES:
Length of hospital stay. | Lead-in phase visit, baseline visit and then at biweekly visits until discharge, an expected average period from lead-in to discharge of seven weeks.
  Firstly, compare the length of hospitalization between study arms. Secondly, measure plasma proline levels and peripheral gene expression, and examine the relationship via regression modeling, with the length of hospitalization.
Number of participants with adverse events as a measure of safety. | Throughout 10 week treatment study period.
  To evaluate the safety of vitamin D supplementation for schizophrenic or schizoaffective patients, by collecting data on all adverse events.
Clinical response to supplementation with vitamin D. | Baseline (start of vitamin D supplementation) through ten weeks of treatment.
  To evaluate a clinical response to vitamin D supplementation by the change in the Brief Ratings Psychiatric Scale.
Clinical response to supplementation with vitamin D. | Baseline (start of vitamin D supplementation) through ten weeks of treatment.
  To evaluate a clinical response to vitamin D supplementation by the change in the Wechsler Adult Intelligence scale.
Clinical response to supplementation with vitamin D. | Baseline (start of vitamin D supplementation) through ten weeks of treatment.
  To evaluate a clinical response to vitamin D supplementation by the change in the Clinical Global Impression scale.

CONTACTS AND LOCATIONS:
Overall Officials: James D Clelland, Principal Investigator — NYU Langone Health
Locations (1):
- Bellevue Hospital Center, New York, New York, United States